CLINICAL TRIAL: NCT05215704
Title: Ex Vivo Characterization and Targeting of the Latent HIV Infected Reservoir to Cure HIV
Acronym: EX VIVO
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Casper Rokx, Principal Investigator, Erasmus Medical Center
Other Study IDs: NL42819.078.12
Record Dates: First submitted 2021-12-15; First posted 2022-01-31 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: HIV Infections; HIV-1-infection; HIV-2 Infection
Keywords: HIV; HIV cure; HIV reservoir
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and leucapheresis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Combination antiretroviral therapy (cART) blocks intracellular human immunodeficiency virus (HIV) replication in CD4+ T-lymphocytes, but fails to eliminate latent HIV infected CD4+ T-lymphocytes. About 7 (range <1-100) in 106 of these cells are latently infected and can cause reactivation of proviral HIV when cART is stopped. These latently infected cells form the reservoir and must be targeted in order to cure HIV. We would like to further investigate this reservoir and assess potential interventions to eradicate it. One promising option is to further study the influence of HIV latency disruptors (latency reversing agents, LRA) on the HIV infected reservoir. These agents are used in shock and kill strategies that disrupt latency by LRA followed by the selective (induced) killing of the reservoir cell due to viro-pathogenic effects.

For accurate assessment of the reservoir and potential cure strategies, including the impact of LRA on the reservoir, a large reservoir and sufficient cells for analysis are desirable. Our understanding on the reservoir comes from in vitro lymphocyte models and early ex vivo studies. Additional studies of patients with different clinical phenotypes including untreated versus treated versus the rare individuals that control HIV spontaneously are increasingly relevant to the field. Especially this last category represent biological examples of viral control without cART and are useful to study the factors that set them apart from those that need treatment for their HIV. This study aims to deepen our understanding of the HIV reservoir and cure strategies, foremost, shock and kill strategies. We will do this by setting up a durable ex vivo platform for HIV reservoir and cure studies of which the samples can be used for hypothesis generation for in-vivo studies.

A project from the Erasmus MC HIV Eradication Group (EHEG).

DETAILED DESCRIPTION:
This is a prospective cross-sectional cohort study used for ex vivo studies using material from HIV infected individuals. Peripheral blood mononuclear cells (PBMC's) and whole blood are obtained through leukapheresis and blood sampling at a single timepoint. Relevant clinical data will be collected to support interpretation of ex vivo experimental results. In vitro experiments are performed on patient derived material. In a substudy, patients can consent to longitudinal follow up with yearly sampling for 4 years.

Reservoir characteristics and efficacy of shock and kill strategies as defined in the endpoints will be explored between patients with different HIV clinical phenotypes. This allows us to identify discriminative factors useful to develop future cure strategies in clinic. We will therefore aim to include the following patients groups in the cohort:

* HIV-1 patients including B and non-B subtypes patients
* HIV-2 patients
* Long term non progressors (plasma HIV-RNA <2000c/mL without cART)
* Elite controllers (plasma HIV-RNA <50c/mL without cART)
* Post-treatment controller (plasma HIV-RNA <2000c/mL after permanent cART interruption)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Confirmed HIV-1 or HIV-2 infection.

Exclusion Criteria:

1. Inability to place 2.5 cm venous catheter or perform phlebotomy
2. Major comorbidities:

   A. Severe symptomatic anemia B. Recent symptomatic cardiovascular event (unstable angina pectoris, decompensated heart failure, myocardial infarction).
3. The inability to participate due to any other relevant medical, social, environmental, psychological, factors or according to the HIV treating physician's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Otherwise healthy adult HIV infected patients will be recruited at the Erasmus MC outpatient clinic of infectious diseases
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of HIV patients with a measurable proviral reservoir measured by molecular, flowcytometric and culture based assays | 10-15 years

SECONDARY OUTCOMES:
The level of reactivation of latently HIV infected PBMCs after treatment ex vivo with established and novel HIV cure compounds (alone and in combination) as assessed by cell-associated HIVRNA. | 10-15 years
The HIV reservoir size and activity as assessed by molecular, flowcytometric, and culture based assays ex vivo. | 10-15 years
The HIV reservoir susceptibility to shock and kill strategies as assessed by molecular, flowcytometric, and culture based assays. | 10-15 years
The HIV reservoir size, activity, and susceptibility to shock and kill strategies in relation to clinical phenotypes. | 10-15 years
To measure predictive biomarkers of the size and activity of the latent HIV reservoir as assessed by molecular, flowcytometric and culture based assay ex vivo. | 10-15 years
The number of newly setup assays that measure the size of the proviral reservoir and are validated with current established molecular, flowcytometric and culture based assays. | 10-15 years

CONTACTS AND LOCATIONS:
Overall Officials: Casper Rokx, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Centre, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided